CLINICAL TRIAL: NCT03724734
Title: A Double-blind, Cross-over Comparison of Closed Loop Versus Conventional Deep Brain Stimulation of the Subthalamic Nucleus in the Treatment of Parkinson's Disease
Brief Title: Trial of Adaptive Deep Brain Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. George's Hospital, London (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Erlick AC Pereira DM FRCS, Senior Lecturer in Neurosurgery, St. George's Hospital, London
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 256068
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease
Keywords: subthalamic nucleus; deep brain stimulation; closed-loop
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Patients will be randomised as to whether they receive conventional DBS or adaptive DBS first. Thereafter they will cross-over to the second type of stimulation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be told which form of stimulation is being applied and the main measures used to evaluate the outcome of the study will be video-taped performance on a number of motor tasks and the video-taping of mobility during arousals and awakenings from sleep.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive DBS (Experimental): We will use our custom-built externalized research system (ERS) to deliver adaptive stimulation to the subthalamic nuclei.
  Interventions: Device: Adaptive DBS
- Conventional DBS (Active Comparator): We will use our custom-built externalized research system (ERS) to deliver continuous stimulation to the subthalamic nuclei.
  Interventions: Device: Conventional DBS

INTERVENTIONS:
Device: Adaptive DBS — We will use our custom-built externalized research system (ERS) to allow recordings and stimulation. The device is small and lightweight and communicates wirelessly with a personal computer. The electrical connections to the DBS leads will be through temporary extensions with appropriate mechanical slack. To allow for stimulation return, a conductive clip to the ERS case will be connected to a conducting (ECG) pad placed over chest. Periodic impedance checks will ensure this connection is robust through the course of the experiment. The patient can be ambulant whilst wearing the device.
  Arms: Adaptive DBS
Device: Conventional DBS — We will use our custom-built externalized research system (ERS) to deliver continuous conventional stimulation.
  Arms: Conventional DBS

SUMMARY:
Currently, treatment of Parkinson's Disease with deep brain stimulation (DBS) uses continuous high frequency stimulation. The investigators have previously shown that by controlling the stimulation using feedback from the brain and only delivering stimulation when needed side-effects like speech disturbance can be reduced. Here the investigators contrast conventional DBS with adaptive DBS while patients are awake and sleeping.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the major neurological movement disorder in terms of both prevalence and morbidity, and in associated health care and social care costs. In the United Kingdom about 120,000 people are affected and associated costs are estimated at £ 2 billion per year. The current gold standard treatment for PD is levodopa therapy, however its use is limited by the development of motor complications in up to 80% of patients over a 5-10 year period. This has led to a resurgence in functional neurosurgery for PD over the last three decades.

Deep brain stimulation (DBS) is now accepted treatment for patients with severe PD and is supported by the Food and Drug Administration in the USA and National Institute of Clinical Excellence in the UK with trials providing evidence that it improves quality of life over best medical treatment. However, due to partial efficacy and side effects its potential is relatively limited and it has so far generally been restricted to patients with severe disease and uncontrollable motor complications with medical therapy.

Currently DBS provides continuous and fixed stimulation, but this constant stimulation promotes side-effects like speech disturbance. Research by the investigators has shown that by controlling the stimulation and only delivering it when needed side-effects can be reduced. To show this the investigators developed a form of adaptive DBS in which they controlled how much stimulation is delivered by directly recording the brain's activity from the electrode used for brain stimulation. This provides a feedback signal.

However, although adaptive DBS works in an acute research setting, there are still several questions to be answered before it can be translated in to a durable therapy option. The main remaining questions are whether the amelioration of Parkinsonian symptoms is maintained over periods longer than an hour or so, and whether it is triggered when arousals occur during sleep. The latter is important to ensure that mobility is maintained when turning in bed and during bathroom visits.

The Investigators would like to contrast conventional (continuous) DBS with adaptive DBS when the same patients with Parkinsons are treated while both awake and asleep. Thus they can follow treatment effects during the day and at night, in sleep. Patients will receive the two types of stimulation in randomised order. Patients will not be told which form of stimulation is being applied and the main measures used to evaluate the outcome of the study will be video-taped performance on a number of motor tasks and the video-taping of mobility during arousals and awakenings from sleep. Assessment of video-tapes is desirable as assessors can then be blind to the treatment being applied. Thus assessments should not be biased.

Patients will undergo our standard 2-part DBS implantation. The experiments will be performed whilst the patients are inpatients between the two operations and will therefore not require any extra procedures, extra hospital stay or incur delay in starting therapeutic DBS.

The DBS electrode has four contacts, and the electrodes are bilaterally implanted. Patients will be requested to withhold their usual medication overnight so that they are first assessed off medication on each morning. Each morning we will start with some screening. On the first of day this will involve finding the best contact for adaptive stimulation on the DBS electrode on the two sides. DBS stimulation will be evaluated in order to find the best contact, voltage and stimulation settings for each individual patient. This assessment is similar to the standard clinical procedure experienced by patients when seen as outpatients following surgery. The investigators will confirm that the settings remain appropriate during the morning screening on the next day.

The investigators will use our custom-built externalized research system (ERS) to allow recordings and stimulation. The ERS will be affixed to the subject with sticky tape or a bandage. The device is small and lightweight and communicates with a personal computer. The electrical connections to the DBS leads will be through temporary extensions with appropriate mechanical slack. The temporary extensions will be later replaced at stimulator implant with new sterile extensions. To allow for stimulation return, a conductive clip to the ERS case will be connected to a conducting (ECG) pad placed over chest. Periodic impedance checks will ensure this connection is robust through the course of the experiment. The patient can be ambulant whilst wearing the device. The safety of the ERS will be reviewed independently prior to the start of the study.

Patients will be randomised as to whether they receive conventional DBS or adaptive DBS and will then cross-over to the second type of stimulation. All procedures will be repeated in matched form in the two treatment periods. The patient's usual medication will be started once each screening test is completed and the medication continued through-out the day.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be patients undergoing DBS of the subthalamic nucleus for the treatment of severe Parkinson's disease. Severe Parkinson's disease is defined as marked motor fluctuations (off periods and dyskinesias) despite optimal medical management. This is determined by the patient's clinical team.
* Able to give consent.

Exclusion Criteria:

* Cognitive impairment (judged by the clinician taking consent as not having sufficient mental capacity to understand the study and its requirements). This includes anyone who, in the opinion of the clinician taking consent, is unlikely to retain sufficient mental capacity for the duration of their involvement in the study.
* Intracranial bleeding, confusion, cerebrospinal fluid leak or any other complication after the first stage of surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Daytime Assessment | 1 day
  Average of blinded videoed United Parkinson's Disease Rating Scale motor score repeated every 3 hours through the day. Score range 0-108. Higher score is worse outcome.
Night time assessment | 1 night
  Average blinded videoed assessment scores of mobility during sleep arousals and awakenings. Score range 0-10. Higher score is worse outcome.

SECONDARY OUTCOMES:
Energy delivered | 1 day/night cycle
  Power consumption (total electrical energy delivered, TEED, over 24h). Measure not bounded. Higher values are worse outcome.
Tremor severity | 1 day/night cycle
  Average accelerometer tremor-band power from limb most affected by tremor. Measure not bounded. Higher values are worse outcome.
Objective motor impairment | 1 day
  Average of timed finger tapping repeated every 3 hours through the day. Measure not bounded. Higher values are better outcome.
Speech impairment | 1 day
  Average of blinded Speech Intelligibility Test score repeated every 3 hours through the day. Scale 0-100. Higher values are better outcome.
Dyskinesia severity | 1 day
  Average of blinded Part 3 of United Dyskinesia Rating Scale score repeated every 3 hours through the day. Rating scale from 0-55. Higher scores are worse impairment.
Sleep quality: score | 1 night
  Sleep quality scale score. 10 point scale. High score is better outcome.
Power efficiency | 1 day
  Power efficiency (mean United Parkinson's Disease Rating Scale motor score divided by the total electrical energy delivered per 24 hours). Measure is not bounded. Higher values are better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Erlick Pereira, DM FRCS, Principal Investigator — St George's University Hospital

IPD SHARING:
Plan to Share IPD: No